CLINICAL TRIAL: NCT04360876
Title: Targeted Steroids for ARDS Due to COVID-19 Pneumonia: A Pilot Randomized Clinical Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding not received
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0811
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: COVID-19; ARDS
Keywords: Corticosteroids; Dexamethasone; COVID-19 Pneumonia; ARDS
MeSH Terms: conditions — COVID-19 | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Single-center, Phase 2a, pragmatic, randomized, double-blinded, placebo-controlled
Who Masked: Participant, Care Provider
Masking Description: Participants confirmed to meet all eligibility criteria who have provided informed consent will be randomized 1:1 to dexamethasone versus placebo. A randomized group assignment will be provided to the investigator or research assistant. Randomization will be performed according to a central randomization scheme and will stratified by site in permuted blocks of varying size.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): Patients assigned to the dexamethasone arm will receive an intravenous dose of 20 mg once daily from day 1 to day 5 which will be reduced to 10mg once daily from day 6 to day 10. Intravenous infusion bags divided into 10 doses will be provided at randomization by the investigational pharmacy. The time from randomization to time for first medication administration will be 4 hours or less. All infusions - dexamethasone and placebo - will be manufactured by the investigational pharmacy at the University of Colorado.
  Interventions: Drug: Dexamethasone injection
- Placebo (Placebo Comparator): Participants randomized to the control group will received placebo intravenously for 10 days, one dose per day. Intravenous infusion bags divided into 10 doses will be provided at randomization by the investigational pharmacy. The placebo infusion bags will be as similar as possible to the dexamethasone infusion bags to ensure blinding.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dexamethasone injection — Dexamethasone intravenous 20mg daily for 5 days followed by 10mg daily for 5 days
  Arms: Dexamethasone
Drug: Placebos — Placebo delivered intravenously on the same dosing schedule as dexamethasone
  Arms: Placebo

SUMMARY:
This trial will determine the safety and estimate efficacy of targeted corticosteroids in mechanically ventilated patients with the hyper-inflammatory sub phenotype of ARDS due to coronavirus disease 2019 (COVID-19) by implementing a Phase 2A clinical trial.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a common, life-threatening pulmonary process which frequently requires mechanical ventilation and has a hospital mortality as high as 40%. No specific pharmacologic therapy has proven efficacy to treat ARDS. Corticosteroids have been investigated as a treatment for ARDS with conflicting results. Two sub phenotypes of ARDS have been described. One is hypo-inflammatory, associated with lower levels of circulating cytokines and therefore greater ventilator free days and a lower mortality. The second sub-phenotype is hyper-inflammatory with elevated cytokine levels, elevated acute phase reactants such as ferritin and c-reactive protein (CRP).

Many patients infected with the novel Coronavirus (SARS-CoV-2), the causative agent of CVOID-19, present with an exaggerated inflammatory response which leads to the hyper-inflammatory sub-phenotype of ARDS. These patients may derive great benefit from corticosteroids. Accordingly,this study will determine the safety and estimate efficacy of targeted corticosteroids in mechanically ventilated patients with the hyper-inflammatory sub phenotype of ARDS due to COVID-19

Hypothesis: Early administration of dexamethasone to patients with the hyper-inflammatory sub-phenotype of ARDS due to COVID-19 pneumonia is a safe intervention which increases ventilator free days

Approach: This is a single-center, phase 2a, pragmatic, randomized, double-blinded, placebo-controlled study accessing the safety and efficacy of dexamethasone for mechanically ventilated patients with ARDS due to COVID-19 infection. Primary outcome will be ventilator free days at day 28.

Understanding the safety and efficacy of corticosteroids in ARDS due to COVID-19 pneumonia could have dramatic implications for critically ill patients. Patients who present with an ARDS sub-type characterized by exaggerated inflammation may particularly benefit from this intervention. Corticosteroids may represent a simple and safe treatment for patients with the most severe form of COVID-19 infection and has the potential to save thousands of lives.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female Adult ≥ 18 years of age at time of enrollment
2. Laboratory confirmed SARS-CoV-2 infection determined by PCR within 14 days prior to randomization and no alternative explanation for current clinical condition
3. Moderate or Severe ARDS (PaO2:FiO2 ratio ≤ 200mmHg) requiring mechanical ventilation within 7 days prior to randomization
4. Hyper-inflammatory ARDS Sub-Phenotype defined as any one of the following:

   1. C-Reactive Protein (CRP) > 100mg/dL
   2. D-Dimer > 600ng/mL
   3. IL-6 > 10pg/mL
5. Willing and/or able to comply with study-related procedures and assessments
6. Provide informed consent signed by study patient or legally acceptable representative

Exclusion Criteria:

1. Age < 18 years
2. In the opinion of the investigator, not expected to survive for more than 48 hours from screening
3. Presence of any of the following abnormal laboratory values at screening

   1. Absolute neutrophil count (ANC) < 2,000mm3
   2. Alanine Transferase (ALT) or Aspartate Transferase (AST) > 5 times upper limit of normal
4. Use of systemic corticosteroid therapy within 7 days of study enrollment
5. Known or suspected active bacterial, fungal or mycobacterial infections including tuberculosis (TB)
6. Participation in a double-blind clinical research study evaluating an investigational product or therapy within 3 months and less than 5 half-lives of investigational product prior to the screening visit. Exception: The use of remdesivir, hydroxychloroquine, or other treatments being used for COVID-19 infection in the context of an open-label study or compassionate use protocol is permitted
7. Any physical examination findings, and/or history of any illness, concomitant medication or recent live vaccines that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study
8. Prisoner
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Ventilator Free Days (VFD) at Day 28 | 28 Days
  Total number of ventilator free days to day 28 of hospitalization. If a patient dies prior to day 28, they will be counted as zero ventilator free days. Follow up will be performed via phone or electronically to determine ventilator free status of those patients discharged prior to day 28.

SECONDARY OUTCOMES:
Clinical Status at day 14 as measured by World Health Organization (WHO) 7-point ordinal scale. | 14 Days
  1. Not hospitalized, no limitations on activities; 2. Not hospitalized, limitation on activities; 3. Hospitalized, not requiring supplemental oxygen; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 6. Hospitalized, on invasive mechanical ventilation or ECMO; 7. Death.
Clinical Status at day 28 as measured by WHO 7-point ordinal scale | 28 Days
In-Hospital Mortality at day 28 | 28 Days
In-Hospital Mortality at day 90 | 90 Days
Time to Mortality to day 28 | 28 Days
ICU-free days to day 28 | 28 Days
Hospital Length of Stay among survivors to day 90 | 90 Days
Severity of ARDS to day 10 | 10 Days
Days to resolution of fever | 28 Days
Change in C-Reactive Protein (CRP) level from baseline to day 10 | 10 Days
Vasopressor-free days to day 28 | 28 Days
Renal replacement-free days to day 28 | 28 Days
Duration of mechanical ventilation to day 28 | 28 Days
Oxygenation-free days to day 28 | 28 Days
Incidence of New Mechanical Ventilation to day 28 | 28 Days
Change in sequential organ failure assessment (SOFA) score from baseline to day 10 | 10 Days
In-hospital adverse events to day 28 | 28 Days
Discontinuation of study drug infusion | 10 Days

IPD SHARING:
Plan to Share IPD: No
No Plan